CLINICAL TRIAL: NCT01069146
Title: Mild Therapeutic Hypothermia During Severe Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Pr Erwan L'HER, MD, PhD, CHU Brest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hymosh
Record Dates: First submitted 2010-02-13; First posted 2010-02-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Sepsis
Keywords: sepsis,; septic shock,; therapeutic hypothermia
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mild therapeutic hypothermia (Experimental): Sepsis treatment according to standard guidelines plus mild therapeutic hypothermia
  Interventions: Procedure: Mild therapeutic hypothermia induction
- Control (No Intervention): Sepsis treatment according to standard guidelines

INTERVENTIONS:
Procedure: Mild therapeutic hypothermia induction — Mild Therapeutic hypothermia was induced immediately after patient inclusion. Patients were cooled between 32 and 34°c (33 ± 1°C; 90 and 93°F) for 36 hours, using the automatic mode of an external water cooling blanket (Meditherm II®, Gaymar, Orchard Park, NY, USA). The machine constantly compares actual patient temperature (measured by a rectal probe) with the set point, and automatically adjusts the blanket water temperature so that the desired patient temperature is achieved. The target temperature was to be reached within eight hour following inclusion. Rewarming was only passive (blanket switched off), and paralytic agents were to be stopped when the body temperature reached back 36°C (97°F).
  Arms: Mild therapeutic hypothermia

SUMMARY:
Objectives: to evaluate the feasibility, the safety and the effects on physiological parameters of mild therapeutic hypothermia during septic shock.

Design: a randomized, controlled, pilot physiological study. Setting: a 15-beds university-affiliated intensive care unit of a teaching Hospital.

Patients: twenty ventilated and sedated adults patients with septic shock Intervention: Mild therapeutic hypothermia between 32 and 34°C during 36 consecutive hours using an external water cooling blanket.

ELIGIBILITY:
Inclusion Criteria:

* age > 18-yrs,
* sedation and mechanical ventilation for at least 48-hrs,
* the diagnosis of septic shock according to standard guidelines.

Exclusion Criteria:

* bradycardia < 50 bpm, or any severe ventricular rhythm disturbances,
* pregnancy,
* need for emergent surgery or any other complementary exam involving patient transport within the sixth hours following inclusion,
* decision to withdraw or withhold life support,
* predictable death within six hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
feasibility of hypothermia induction during sepsis | 48 hours

SECONDARY OUTCOMES:
hemodynamic parameters evolution | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Réanimation Médicale, CHU de la Cavale Blanche, Brest, France